CLINICAL TRIAL: NCT03290326
Title: Feasibility and Safety of a High-Frequency Transcranial Alternating Current Stimulation Intervention for Amyloid-β Reduction in Alzheimer's Disease
Brief Title: tACS for Amyloid-β Reduction in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Emiliano Santarnecchi, Associate Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000373
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Memory Problems
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tACS (Experimental): Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) will be applied for 1 hour in 10 sessions on consecutive weekdays. The tACS intervention (10 sessions) will be preceded and followed by amyloid PET imaging as well as a clinical/cognitive evaluation. The assessment of adverse effects will constitute a Primary outcome measure. Changes in amyloid load in the stimulated brain region will be evaluated and constitute a secondary outcome of the study. Clinically relevant changes in cognitive and clinical scores will be also evaluated as secondary outcomes. Stimulation will be also preceded and followed by electroencephalography (EEG) recording aimed at assessing changes in spectral power in the gamma band.
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — tACS will be applied at a frequency of 40Hz and targeting the area of maximal tracer uptake on amyloid PET imaging using an individualized multielectrode design to maximize the induced electrical current to the target region.

SUMMARY:
Alzheimer's Disease (AD) is characterized by amyloid-β (Aβ) plaque buildup and phosphorylated tau (p-tau) in the brain, as well as widespread neurodegeneration. The evidence suggests that both amyloid and tau play a critical role in AD and interventions that reliably and safely decrease the intracerebral burden of amyloid or tau could potentially be of marked clinical importance. Currently, therapeutic options are very limited and while there are pharmacologic interventions that transiently improve cognitive function, there are no treatments that alter disease progression. The current study seeks to use a novel therapeutic intervention that uses noninvasive brain stimulation to target amyloid in the brain. The investigators anticipate this will decrease the amyloid levels in the brain, as evidence by Positron Emission Tomography (PET) imaging.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is characterized by amyloid-β (Aβ) plaque buildup and phosphorylated tau (p-tau) in the brain, as well as widespread neurodegeneration. There is no current treatments that alter disease progression.

Investigators will recruit 20 individuals with AD with evidence of amyloid placques in the brain through Positron Emission Tomography (PET) imaging. Investigators will use a novel approach, transcranial alternating current stimulation (tACS), to target the region of maximum amyloid burden in the brain. All participants will receive tACS. Each individual's participation in the study will consist of approximately 16 visits: 3 days for screening/baseline procedures as described below, 10 tACS study visits, and 3 days for follow-up assessments. Subjects will undergo baseline cognitive assessment, structural and functional MRI characterization, and resting-state EEG measurement. Additionally, patients will undergo a tACS-EEG recording session to assess brain plasticity levels and identify markers of response to stimulation. All subjects will then undergo 10 1-hour sessions of gamma-frequency (40 Hz) tACS, targeted to the region of maximal tracer uptake on the amyloid PET study. Subjects will take a standardized adverse effect questionnaire before and after each session and complete a short cognitive test after each session to demonstrate safety and tolerability. At the end of the 10 sessions, subjects will then repeat the baseline assessments, followed by repeat amyloid PET imaging to assess for changes in amyloid burden.

Investigators anticipate that targeting the region of amyloid burden in the brain with tACS will reduce the amyloid burden as evidence by the follow up PET imaging and show improvement on electrophysiological measures of brain function and on cognitive testing. If our prediction is correct, this will will provide a critical first step in the development of a novel intervention to prevent and treat AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of mild AD defined by: Clinical Dementia Rating (CDR) = 0.5-1, Mini Mental State Examination (MMSE) >/= 20, Demonstration or history of memory impairments
* Amyloid positive PET imaging
* At least 45 years old
* On a stable dose of medications for memory loss including cholinesterase inhibitors (e.g. donepezil, rivastigmine or memantine) as defined as 6 consecutive weeks of treatment at an unchanging dose
* Intelligence Quotient (IQ) > 85 as determined by the Wechsler Test of Adult Reading (WTAR) and no history of intellectual disability

Exclusion Criteria:

* Current history of poorly controlled migraines including chronic medication for migraine prevention
* Current or past history of any neurological disorder other than dementia, such as epilepsy, stroke, progressive neurologic disease (e.g. multiple sclerosis) or intracranial brain lesions; and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment.
* Past or current history of major depression, bipolar disorder or psychotic disorders, or any other major psychiatric condition.
* Contraindication for undergoing MRI or receiving Transcranial Magnetic Stimulation (TMS) or tACS,

  • History of fainting spells of unknown or undetermined etiology that might constitute seizures.
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or immediate (1st degree relative) family history of epilepsy; with the exception of a single seizure of benign etiology (e.g. febrile seizure) in the judgment of the investigator.
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.).
* Metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, Transcutaneous Electrical Nerve Stimulator (TENS) unit, ventriculo-peritoneal shunt, cochlear implant, unless cleared by the study MD.
* Substance abuse or dependence within the past six months.
* Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination of Central Nervous System (CNS) active drugs.
* All female participants that are pre-menopausal will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study.
* BMI > 40 kg/m2. We will limit the BMI to <40 kg/m2 because of weight limits of the scanner bed and width limits of the MRI.
* Subjects who, in the investigator's opinion, might not be suitable for the study
* A hair style or head dress that prevents electrode contact with the scalp or would interfere with the stimulation (for example: thick braids, hair weave, afro, wig)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Santarnecchi, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sprugnoli G, Munsch F, Cappon D, Paciorek R, Macone J, Connor A, El Fakhri G, Salvador R, Ruffini G, Donohoe K, Shafi MM, Press D, Alsop DC, Pascual Leone A, Santarnecchi E. Impact of multisession 40Hz tACS on hippocampal perfusion in patients with Alzheimer's disease. Alzheimers Res Ther. 2021 Dec 20;13(1):203. doi: 10.1186/s13195-021-00922-4. PMID 34930421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 17 enrolled participants, 10 met inclusion criteria and underwent transcranial alternating current stimulation (tACS)
Pre-assignment Details: During the screening and baseline procedures 7 participants screened out for the following reasons: 4 participants screened out on cognitive testing measures, being either too advanced or too mild, 2 participants did not meet 6 weeks stable medication inclusion criteria, and 1 participant screened out due to incidental findings on the baseline MRI
Groups:
- tACS: Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) was applied for 1 hour in 10 sessions on consecutive weekdays.
Period: Overall Study
Arm/Group | tACS
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | tACS
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  Age: 55 | 1
  Age: 57 | 1
  Age: 63 | 1
  Age: 75 | 1
  Age: 76 | 2
  Age: 78 | 2
  Age: 79 | 1
  Age: 83 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Amyloid Burden
Description: Changes in the amyloid load observed via PET imaging will be evaluated by comparing PET data acquired before and after the 10 tACS sessions. The metric used is SUVR, a measure of the amount of proteins in the brain identified at the PET exam. We will calculate the difference between pre and post tACS SUVR (dSUVR) for the entire brain and report the average value (and standard deviation) for the entire group of patients. A negative value express a decrease in the amount of proteins in the brain post tACS intervention. It must be considered that dSUVR values refer to the entire brain, however patients were treated according to personalized tACS montages targeting patient-specific regions mostly affected by the pathology. This might have led to slightly different changes in SUVR in different part of the brain across participants. Also, as per standard procedures, results are presented at group level, i.e. without considering individual differences in longitudinal amyloid load changes.
Time Frame: Up to six weeks
Population: Mild to Moderate Alzheimer's Disease patients
Measure: Mean (Standard Deviation); unit: dSUVR
Groups:
- tACS: Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) will be applied for 1 hour in 10 sessions on consecutive weekdays. The tACS intervention (10 sessions) will be preceded and followed by amyloid PET imaging as well as a clinical/cognitive evaluation. The assessment of adverse effects will constitute a Primary outcome measure. Changes in amyloid load in the stimulated brain region will be evaluated and constitute a secondary outcome of the study. Clinically relevant changes in cognitive and clinical scores will be also evaluated as secondary outcomes. Stimulation will be also preceded and followed by electroencephalography (EEG) recording aimed at assessing changes in spectral power in the gamma band.
  tACS will be applied at a frequency of 40Hz and targeting the area of maximal tracer uptake on amyloid PET imaging using an individualized multielectrode design to maximize the induced electrical current to the target region.
Arm/Group | tACS
Number analyzed (Participants) | 10
dSUVR | -1.55 (0.9)

2. Secondary Outcome: Change in EEG Gamma-band Spectral Power
Description: EEG power spectral densities (PSD) before and after the tACS intervention were evaluated, specifically absolute and relative power density values (μV2/Hz) were calculated within the gamma band (35-45Hz). Changes in the spectral power are reported in term of percentage of changes in relative spectral power from Pre to Post tACS intervention.
Time Frame: Up to six weeks
Population: The assessment of the effect of 40 Hz tACS on EEG gamma-band spectral power.
Measure: Mean (Standard Deviation); unit: % difference in spectral power (μV2/Hz)
Groups:
- tACS 40Hz: Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) will be applied for 1 hour in 10 sessions on consecutive weekdays. The tACS intervention (10 sessions) will be preceded and followed by amyloid, microglia and tau PET imaging as well as a clinical/cognitive evaluation. The assessment of the effect of stimulation on microglia activation, amyloid deposition and tau deposition will constitute a primary outcome measure. Assessment of adverse effects will be also evaluated as a secondary outcome. The effect of brain stimulation on brain connectivity will be assessed by EEG and cognitive function.
  Transcranial Alternating Current Stimulation (tACS): tACS will be applied at a frequency of 40Hz and targeting the area of maximal tracer uptake on amyloid PET imaging using an individualized multielectrode design to maximize the induced electrical current to the target region.
Arm/Group | tACS 40Hz
Number analyzed (Participants) | 10
% difference in spectral power (μV2/Hz) | 23.5 (13.4)
Statistical Analysis 1: Comparison: tACS 40Hz; One-way ANOVA was conducted to compare the effect of 40Hz tACS on EEG gamma-band spectral power. Power changes were expressed as percentage relative power variations, accordingly with the event-related synchronization/desynchronization (ERS/ERD) index; Test type: Other; p < 0.01, ANOVA

3. Secondary Outcome: Change in Adas-Cog Score
Description: Change in Adas-Cog score will be reported, to document a potential clinical benefit of tACS. The scale ranges from a total score of 0-70 with higher score indicating greater cognitive impairment.
Time Frame: Up to six weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- tACS: Transcranial alternating current stimulation (tACS) tuned at the frequency of 40Hz (gamma frequency) will be applied for 1 hour in 10 sessions on consecutive weekdays.
Arm/Group | tACS
Number analyzed (Participants) | 10
Scores on a scale | -0.97 (3.88)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | tACS
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | tACS (N=10)
Headache (General disorders) | 2
Scalp Pain (General disorders) | 2
Neck Pain (General disorders) | 2 — related to TMS positioning
Skin Irritation (General disorders) | 5
Sensations under electrodes (General disorders) | 8 — tingling, burning, itching
Visual Changes (General disorders) | 6 — flashing lights in peripheral vision
Nervousness (General disorders) | 3 — related to cognitive testing
Difficulty concentrating (General disorders) | 2
Hand tingling (General disorders) | 1
Eye pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03290326/Prot_SAP_000.pdf